CLINICAL TRIAL: NCT06634238
Title: INVESTIGATION of the ACUTE EFFECT of MASK USE on WALKING DISTANCE and VITAL SIGNS DURING the INCREMENTAL SHUTTLE WALK TEST in HEALTHY INDIVIDUALS
Brief Title: Acute Mask Effects on Walk Distance and Vital Signs
Status: Not yet recruiting | Type: Observational
Sponsor: Nagihan Acet (Other)
Responsible Party: Sponsor-Investigator, Nagihan Acet, Asst. Prof., Atılım University
Organization: Atılım University (Other)
Other Study IDs: GAZİ UNIVERSİTY
Record Dates: First submitted 2024-10-08; First posted 2024-10-09 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Mask Usage Condition
Keywords: Mask; vital signs; shuttle walk test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Masked Group: Participants who performed the Incremental Shuttle Walk Test (ISWT) while wearing a face mask.
  Interventions: Other: Incremental shuttle walk test
- Unmasked Group: Participants who performed the Incremental Shuttle Walk Test (ISWT) without wearing a face mask.
  Interventions: Other: Incremental shuttle walk test

INTERVENTIONS:
Other: Incremental shuttle walk test — Participants were recommended to wear comfortable clothing and appropriate shoes for the test. To minimize variability, one masked and one unmasked ISWT was performed on the same participant at the same time of day, one day apart

SUMMARY:
The goal of this prospective observational study is to investigate the acute effects of mask use on walking distance and vital signs in healthy individuals aged 18-24 years. The main questions it aims to answer are:

Does wearing a mask affect walking distance during the Incremental Shuttle Walk Test (ISWT)? How does mask use influence heart rate, oxygen saturation, blood pressure, and respiratory rate during the test? Researchers will compare participants performing the ISWT with a mask to those performing it without a mask to determine any differences in walking distance and vital signs.

Participants will:

Complete the ISWT twice: once with a mask and once without a mask, on separate days.

Have their heart rate, oxygen saturation, respiratory rate, blood pressure, and dyspnea perception measured before and after each test.

DETAILED DESCRIPTION:
The incremental shuttle walk test (ISWT) is an exercise test used to evaluate maximum exercise capacity in different chronic diseases. ISWT consists of 12 levels, each lasting 1 minute, where the participant walks back and forth along a 10-meter course. The test involves progressively increasing the pace as the individual moves between two cones placed 9 meters apart. The speed of walking is controlled by an audio signal. Initially, the speed is set at 0.50 m/s and is incremented by 0.17 m/s every minute until reaching a final speed of 2.37 m/s at level 12. The test concludes when the participant is hindered by shortness of breath or reaches a heart rate of 85% of their predicted maximum, or if they cannot sustain the required speed and fail to complete a shuttle for two consecutive attempts. The main result is determined by the distance traveled, which is calculated based on the number of shuttles completed.

The coronavirus pandemic has altered the manner in which routine tests are conducted. Since the beginning of the pandemic, wearing masks in public places has been mandatory, necessitating the use of masks during clinical tests.

There are a limited number of studies on the effects of mask use on the results of exercise tests. In a study investigating the effects of mask use on the results of the 6-minute walk test, no significant difference was found in terms of walking distance, while no significant difference was found in terms of dyspnea perception between the two groups. Similar results were found in another study on this subject.

To the best of our knowledge, there is no study in the literature examining the effect of mask use on the results of the ISWT. The aim of this study is to determine whether there are differences in walking distance, maximal heart rate, oxygen saturation, perception of dyspnea, and respiratory rate between healthy individuals undergoing the ISWT with and without masks.

Individuals aged 18-24 years with a body mass index of less than 30 kg/m² and no known diseases will be included in the study. Individuals who self-report a history of chronic or acute disease/dysfunction that contraindicates or limits participation in exercise testing, those taking prescription medications other than oral contraception, those with known pregnancy status, those using drugs, cigarettes, or alcohol, and those with blood pressure greater than or equal to 160/100 mmHg will be excluded from the study.

Participants will be recommended to wear comfortable clothing and appropriate shoes for the test. To minimize variability, each participant will perform the Incremental Shuttle Walk Test (ISWT) twice, once with a mask and once without a mask, at the same time of day on separate days. Walking distance, respiratory frequency, heart rate, dyspnea perception, and blood pressure will be measured at rest, immediately after the test, and one minute after the test.

Heart rate will be evaluated using a heart rate monitor (Polar FT 100), oxygen saturation will be measured with a portable pulse oximeter, blood pressure will be taken with a sphygmomanometer, respiratory frequency will be measured by counting the number of breaths per minute, and dyspnea perception will be assessed using the Modified Borg Scale.

The Modified Borg Scale is frequently used to evaluate the severity of dyspnea on exertion and at rest. It is a 10-point scale that defines the severity of dyspnea and is known to be a reliable scale for determining dyspnea severity and is related to respiratory function tests.

Statistical analysis will be performed using IBM Statistics SPSS v21.0 (IBM Corp., Armonk, NY, USA). Variables will be assessed using histograms and the Shapiro-Wilk test. For the primary and secondary outcomes, changes in ISWT with and without a mask, the Mann-Whitney U test will be used. Significance will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-24 years.
* Body mass index of less than 30 kg/m².
* No known diseases

Exclusion Criteria:

* Individuals with a self-reported history of chronic or acute disease/dysfunction that contraindicates or limits participation in exercise testing.
* Individuals taking prescription medications other than oral contraception.
* Those with known pregnancy status.
* Individuals who use drugs, cigarettes, or alcohol.
* Individuals with blood pressure greater than ≥160/100 mmHg.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of healthy volunteers, aged between 18 and 24 years, with a body mass index (BMI) of less than 30 kg/m². All participants are free from any known chronic or acute diseases, do not take prescription medications (except for oral contraception), and have no history of drug, alcohol, or cigarette use. Additionally, participants with blood pressure greater than 160/100 mmHg or those with known pregnancy status are excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Heart rate | Before the test and immediately after the test
  Heart rate will be evaluated using a heart rate monitor (Polar FT 100).
Oxygen saturation | Before the test and immediately after the test
  Oxygen saturation will be evaluated with a portable pulse oximeter.
Blood pressure | Before the test and immediately after the test
  Blood pressure will be evaluated by sphygmomanometer.
Respiratory frequency | Before the test and immediately after the test
  Respiratory frequency will be evaluated by counting the number of breaths in a minute, and dyspnea perception was evaluated using the Modified Borg Scale.
Dyspnea perception | Before the test and immediately after the test
  Dyspnea perception will be evaluated using the Modified Borg Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Murat Esmer, Principal Investigator — Gazi University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singh SJ, Morgan MD, Scott S, Walters D, Hardman AE. Development of a shuttle walking test of disability in patients with chronic airways obstruction. Thorax. 1992 Dec;47(12):1019-24. doi: 10.1136/thx.47.12.1019. PMID 1494764
- [Background] Probst VS, Hernandes NA, Teixeira DC, Felcar JM, Mesquita RB, Goncalves CG, Hayashi D, Singh S, Pitta F. Reference values for the incremental shuttle walking test. Respir Med. 2012 Feb;106(2):243-8. doi: 10.1016/j.rmed.2011.07.023. Epub 2011 Aug 23. PMID 21865021
- [Background] Parreira VF, Janaudis-Ferreira T, Evans RA, Mathur S, Goldstein RS, Brooks D. Measurement properties of the incremental shuttle walk test. a systematic review. Chest. 2014 Jun;145(6):1357-1369. doi: 10.1378/chest.13-2071. PMID 24384555
- [Background] Burdon JG, Juniper EF, Killian KJ, Hargreave FE, Campbell EJ. The perception of breathlessness in asthma. Am Rev Respir Dis. 1982 Nov;126(5):825-8. doi: 10.1164/arrd.1982.126.5.825. PMID 7149447
- [Background] Grant S, Aitchison T, Henderson E, Christie J, Zare S, McMurray J, Dargie H. A comparison of the reproducibility and the sensitivity to change of visual analogue scales, Borg scales, and Likert scales in normal subjects during submaximal exercise. Chest. 1999 Nov;116(5):1208-17. doi: 10.1378/chest.116.5.1208. PMID 10559077
- [Background] Wu G, Sanderson B, Bittner V. The 6-minute walk test: how important is the learning effect? Am Heart J. 2003 Jul;146(1):129-33. doi: 10.1016/S0002-8703(03)00119-4. PMID 12851620
- [Background] Goncalves CG, Mesquita R, Hayashi D, Merli MF, Vidotto LS, Fernandes KB, Probst VS. Does the Incremental Shuttle Walking Test require maximal effort in healthy subjects of different ages? Physiotherapy. 2015 Jun;101(2):141-6. doi: 10.1016/j.physio.2014.11.002. Epub 2014 Nov 11. PMID 25700634